CLINICAL TRIAL: NCT00678561
Title: PHASE 2A RANDOMIZED, DOUBLE-BLIND, VEHICLE-CONTROLLED, INTRA-INDIVIDUAL COMPARISON TRIAL ASSESSING SAFETY, TOLERATION, PHARMACOKINETICS AND PILOT EFFICACY OF 4 WEEKS TREATMENT WITH TOPICAL CP-690,550 IN CHRONIC PLAQUE PSORIASIS
Brief Title: Topical CP-690,550 For Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3921038
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Results first posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Psoriasis
Keywords: chronic plaque psoriasis; topical treatment
MeSH Terms: conditions — Psoriasis | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- 2% CP-690,550 QD (Experimental)
  Interventions: Drug: CP-690,550
- 0.2% CP-690,550 QD (Experimental)
  Interventions: Drug: CP-690,550
- 0.02% CP-690,550 QD (Experimental)
  Interventions: Drug: CP-690,550
- 2% CP-690,550 BID (Experimental)
  Interventions: Drug: CP-690,550
- 0.2% CP-690,550 BID (Experimental)
  Interventions: Drug: CP-690,550
- 0.02% CP-690,550 BID (Experimental)
  Interventions: Drug: CP-690,550
- Placebo Vehicle QD (Placebo Comparator)
  Interventions: Drug: Placebo Vehicle
- Placebo Vehicle BID (Placebo Comparator)
  Interventions: Drug: Placebo Vehicle

INTERVENTIONS:
Drug: CP-690,550 — Topical treatment once daily for 28 days
  Arms: 2% CP-690,550 QD
Drug: CP-690,550 — Topical treatment once daily for 28 days
  Arms: 0.2% CP-690,550 QD
Drug: CP-690,550 — Topical treatment once daily for 28 days
  Arms: 0.02% CP-690,550 QD
Drug: CP-690,550 — Topical treatment twice daily for 28 days
  Arms: 2% CP-690,550 BID
Drug: CP-690,550 — Topical treatment twice daily for 28 days
  Arms: 0.2% CP-690,550 BID
Drug: CP-690,550 — Topical treatment twice daily for 28 days
  Arms: 0.02% CP-690,550 BID
Drug: Placebo Vehicle — Topical treatment once daily for 28 days
  Arms: Placebo Vehicle QD
Drug: Placebo Vehicle — Topical treatment twice daily for 28 days
  Arms: Placebo Vehicle BID

SUMMARY:
Study will test effectiveness of an experimental drug applied once or twice daily to two psoriasis plaques. Requires 1 clinic visit each week for 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Having chronic plaque psoriasis for at least 6 months
* Able to withdraw all prior psoriasis treatments
* Must agree to avoid prolonged exposure to the sun and avoid use of tanning booths or other ultraviolet light sources during the study

Exclusion Criteria:

* Evidence of active, latent, or inadequately treated infection with Mycobacterium tuberculosis
* Pregnant or lactating women
* Unwilling to use appropriate contraceptive methods

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2008-10-13 (Actual); Primary Completion 2009-07-09 (Actual); Study Completion 2009-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- United States (14):
  - University of California Irvine, Irvine, California
  - Therapeutics Clinical Research, San Diego, California
  - RUSH University Medical Center, Chicago, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Central Dermatology, PC, St Louis, Missouri
  - Dermatology Consulting Services, High Point, North Carolina
  - The Imaging Center, High Point, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Oregon Medical Research Center, PC, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - DermResearch, Inc., Austin, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
- Canada (6):
  - Guildford Dermatology Specialists, Surrey, British Columbia
  - NewLab Clinical Research Inc., St. John's, Newfoundland and Labrador
  - K.Papp Clinical Research Inc., Waterloo, Ontario
  - Innovaderm Research, Inc., Montreal, Quebec
  - Siena Medical Research, Montreal, Quebec
  - Centre de Recherche Dermatologique du Quebec metropolitain, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Ports WC, Feldman SR, Gupta P, Tan H, Johnson TR, Bissonnette R. Randomized Pilot Clinical Trial of Tofacitinib Solution for Plaque Psoriasis: Challenges of the Intra-Subject Study Design. J Drugs Dermatol. 2015 Aug;14(8):777-84. PMID 26267721
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921038&StudyName=Topical%20CP-690%2C550%20For%20Chronic%20Plaque%20Psoriasis

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the study, enrollment into the 4 once daily dosing regimen treatment groups was discontinued in order to decrease the overall total number of participants to be enrolled.
Groups:
- 2% CP-690,550 Once Daily: CP-690,550 2.0 percent (%) (50 microgram per square centimeter [mcg/cm^2]) gel (active) applied topically on 1 target plaque area, along with matching placebo vehicle on another target plaque area, once daily up to Day 28.
- 0.2% CP-690,550 Once Daily: CP-690,550 0.2% (5 mcg/cm^2), gel (active) applied topically on 1 target plaque area, along with matching placebo vehicle on another target plaque area, once daily up to Day 28.
- 0.02% CP-690,550 Once Daily: CP-690,550 0.02% (0.5 mcg/cm^2) gel (active), applied topically on 1 target plaque area, along with matching placebo vehicle on another target plaque area, once daily up to Day 28.
- Placebo Once Daily: CP-690,550 matching placebo vehicle applied topically on 2 target plaque areas, once daily up to Day 28.
- 2% CP-690,550 Twice Daily: CP-690,550 2.0% (50 mcg/cm^2), gel (active) applied topically on 1 target plaque area, along with matching placebo vehicle on another target plaque area, twice daily up to Day 28.
- 0.2% CP-690,550 Twice Daily: CP-690,550 0.2% (5 mcg/cm^2) gel (active) applied topically on 1 target plaque area, along with matching placebo vehicle on another target plaque area, twice daily up to Day 28.
- 0.02% CP-690,550 Twice Daily: CP-690,550 0.02% (0.5 mcg/cm^2) gel (active) applied topically on 1 target plaque area, along with matching placebo vehicle on another target plaque area, twice daily up to Day 28.
- Placebo Twice Daily: CP-690,550 matching placebo vehicle applied topically on 2 target plaque areas twice daily up to Day 28.
Period: Overall Study
Arm/Group | 2% CP-690,550 Once Daily | 0.2% CP-690,550 Once Daily | 0.02% CP-690,550 Once Daily | Placebo Once Daily | 2% CP-690,550 Twice Daily | 0.2% CP-690,550 Twice Daily | 0.02% CP-690,550 Twice Daily | Placebo Twice Daily
Started | 6 | 6 | 8 | 4 | 17 | 17 | 15 | 8
Completed | 6 | 5 | 7 | 4 | 15 | 16 | 15 | 7
Not Completed | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2% CP-690,550 Once Daily | 0.2% CP-690,550 Once Daily | 0.02% CP-690,550 Once Daily | Placebo Once Daily | 2% CP-690,550 Twice Daily | 0.2% CP-690,550 Twice Daily | 0.02% CP-690,550 Twice Daily | Placebo Twice Daily | Total
Number analyzed (Participants) | 6 | 6 | 8 | 4 | 17 | 17 | 15 | 8 | 81
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.8 (7.3) | 45.7 (11.6) | 50.3 (17.0) | 52.5 (13.1) | 45.9 (10.5) | 43.2 (15.8) | 47.4 (13.0) | 41.1 (17.0) | 46.3 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 1 | 4 | 5 | 2 | 1 | 15
  Male | 5 | 5 | 8 | 3 | 13 | 12 | 13 | 7 | 66

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Target Plaque Severity Score (TPSS) at Week 4
Description: TPSS: all target lesions were scored individually by the investigator for signs of induration, scaling, and erythema. For large target lesions only a portion of the lesion was treated and only the treated portion was rated. Each of the 3 signs was rated on a 5-point severity scale: 0 = none; 1 = slight; 2 = moderate; 3 = marked; 4 = very marked. Total score range for TPSS was 0 to 12, higher score indicated greater severity of disease.
Time Frame: Baseline, Week 4
Population: Full analysis set (FAS) population included all randomized participants who received at least 1 dose of study medication and had a valid baseline with at least one valid post-baseline value for efficacy parameter. N (number of participants analyzed) is signifying those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Percent Change
Groups:
- 0.2% CP-690,550 Once Daily: CP-690,550 0.2% (5 mcg/cm^2) gel (active) applied topically on 1 target plaque area, along with matching placebo vehicle on another target plaque area, once daily up to Day 28.
- Placebo Once Daily: CP-690,550 matching placebo vehicle applied topically on 2 target plaque areas once daily up to Day 28.
- 0.2% CP-690,550 Twice Daily: CP-690,550 0.2% (5 mcg/cm^2) gel applied topically on 1 target plaque area, along with matching placebo gel on another target plaque area, twice daily up to Day 28.
- Placebo Twice Daily: Matching placebo gel applied topically on 2 target plaque areas twice daily up to Day 28.
Arm/Group | 2% CP-690,550 Once Daily | 0.2% CP-690,550 Once Daily | 0.02% CP-690,550 Once Daily | Placebo Once Daily | 2% CP-690,550 Twice Daily | 0.2% CP-690,550 Twice Daily | 0.02% CP-690,550 Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 6 | 6 | 8 | 4 | 15 | 16 | 15 | 7
Percent Change | 2.38 (5.83) | -4.76 (11.66) | 2.48 (11.50) | -4.17 (8.33) | -4.46 (9.23) | -1.77 (20.87) | -3.29 (21.34) | -7.14 (20.11)

2. Secondary Outcome: Percentage of Participants With Success Based on Physician's Global Assessment (PGA) of Target Lesions
Description: PGA of Psoriasis: The investigator scored each target lesion on a 5-point scale, reflecting the erythema, induration and scaling separately for each target lesions. Each parameter was scored from 0 to 4, with appropriate morphologic descriptors. The 5-point scale for PGA was: 0, "clear"; 1, "almost clear"; 2, "mild"; 3, "moderate"; 4 "severe". The sum of the 3 scores was divided by 3 to obtain a final PGA score. Total score range: 0 to 4, higher score indicated greater severity of disease. Success was considered as PGA response of "clear" and "almost clear".
Time Frame: Week 4
Population: FAS population included participants who received at least 1 dose of study medication and had a valid baseline with at least one valid post-baseline value for efficacy assessment. N (number of participants analyzed) is signifying those participants who were evaluable for this measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | 2% CP-690,550 Once Daily | 0.2% CP-690,550 Once Daily | 0.02% CP-690,550 Once Daily | Placebo Once Daily | 2% CP-690,550 Twice Daily | 0.2% CP-690,550 Twice Daily | 0.02% CP-690,550 Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 6 | 6 | 8 | 4 | 15 | 16 | 15 | 7
Percentage of Participants
  Active, Clear | 0.0 | 0.0 | 0.0 | 0.0 | 6.7 | 0.0 | 0.0 | 0.0
  Active, Almost Clear | 0.0 | 0.0 | 0.0 | 0.0 | 13.3 | 25.0 | 33.3 | 14.3
  Vehicle, Clear | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Vehicle, Almost Clear | 0.0 | 0.0 | 0.0 | 0.0 | 26.7 | 25.0 | 13.3 | 0.0

3. Secondary Outcome: Percent Change From Baseline in Target Plaque Severity Score (TPSS) at Week 1, 2 and 3
Description: TPSS: all target lesions were scored individually by the investigator for signs of induration, scaling, and erythema. For large target lesions only a portion of the lesion was treated and only the treated portion was rated. Each of the 3 signs was rated on a 5-point scale: 0 = none; 1 = slight; 2 = moderate; 3 = marked; 4 = very marked. Total score range for TPSS was 0 to 12, higher score indicated greater severity of disease.
Time Frame: Baseline, Week 1, 2, 3
Population: FAS: all randomized participants who received at least 1 dose of study medication; had a valid baseline with at least 1 valid post-baseline efficacy assessment. Here 'N' (number of participants analyzed)= participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | 2% CP-690,550 Once Daily | 0.2% CP-690,550 Once Daily | 0.02% CP-690,550 Once Daily | Placebo Once Daily | 2% CP-690,550 Twice Daily | 0.2% CP-690,550 Twice Daily | 0.02% CP-690,550 Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 6 | 6 | 8 | 4 | 16 | 17 | 15 | 8
percent change
  Week 1 | 0.00 (0.00) | 5.56 (13.61) | -1.39 (9.74) | -16.67 (33.33) | -1.59 (28.97) | 4.24 (16.30) | 2.13 (11.59) | -3.87 (7.19)
  Week 2 | -5.56 (8.61) | 0.93 (8.90) | 0.69 (8.63) | 0.00 (0.00) | -3.49 (16.24) | 0.25 (9.82) | -4.55 (16.11) | -4.42 (13.45)
  Week 3 | 0.00 (0.00) | 2.78 (6.80) | 8.73 (13.52) | -16.67 (28.87) | -4.66 (13.47) | 3.06 (22.74) | -2.99 (16.38) | -2.83 (16.00)

4. Secondary Outcome: Number of Participants With Administration Site Adverse Events
Description: An adverse event was any untoward medical occurrence attributed to study drug in a participant who received study drug. Administration site adverse event included documentation of any clinically significant local reaction, such as erosion, vesicles or scabbing.
Time Frame: Baseline up to 7 to 10 days after last dose of study treatment (maximum up to 38 days)
Population: FAS population included participants who received at least 1 dose of study medication and had a valid baseline with at least one valid post-baseline value for efficacy assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | 2% CP-690,550 Once Daily | 0.2% CP-690,550 Once Daily | 0.02% CP-690,550 Once Daily | Placebo Once Daily | 2% CP-690,550 Twice Daily | 0.2% CP-690,550 Twice Daily | 0.02% CP-690,550 Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 6 | 6 | 8 | 4 | 17 | 17 | 15 | 8
Participants
  Active | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Vehicle | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0

5. Secondary Outcome: Drug Plasma Concentrations of CP-690,555
Description: Concentrations below the limit of quantification (LOQ) were not estimable. The LOQ was 0.1 ng/mL.
Time Frame: 0 hour (pre-dose) on Day 14 and 0 hour (pre-dose), 1, 2, 9 hours post-dose on Day 28
Population: FAS: all randomized participants who received at least 1 dose of study medication; had a valid baseline with at least 1 valid post-baseline efficacy assessment of CP-690,550. Participants of reporting groups 2%, 0.2% and 0.02% CP-690,550 Once Daily regimen had no post-baseline measurable concentration of CP-690,550. "Overall number of participants analyzed" = who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 2% CP-690,550 Twice Daily | 0.2% CP-690,550 Twice Daily | 0.02% CP-690,550 Twice Daily
Number analyzed (Participants) | 3 | 2 | 1
nanogram per milliliter (ng/mL)
  0 hour post-dose | 0.183 (0.054) | 0.116 (0.020) | NA (NA) — Mean and standard deviation were not estimable as data was below LOQ.
  1 hour post-dose | 0.174 (0.046) | NA (NA) — Mean and standard deviation were not estimable as data was below LOQ. | 0.126 (NA) — Standard deviation not calculated as only 1 participant was evaluable.
  2 hour post-dose | 0.191 (0.059) | NA (NA) — Mean and standard deviation were not estimable as data was below LOQ. | 0.115 (NA) — Standard deviation not calculated as only 1 participant was evaluable.
  9 hour post-dose | 0.160 (0.039) | NA (NA) — Mean and standard deviation were not estimable as data was below LOQ. | 0.102 (NA) — Standard deviation not calculated as only 1 participant was evaluable.

6. Secondary Outcome: Skin Biopsy Drug Concentrations
Description: Skin biopsy drug concentrations was measured via drug levels in dermis and expressed as nanogram of drug per milligram (mg) of dermis weight. Tissue concentration (ng/mg) = (ng drug/mL extraction solvent multiplied by mL extraction solvent) divided by mg tissue weight; 1 mL of extraction solvent was used.
Time Frame: Day 28
Population: FAS population included participants who received at least 1 dose of study medication and had a valid baseline with at least one valid post-baseline value for efficacy assessment. Overall number of participants analyzed = participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: ng/mg
Arm/Group | 2% CP-690,550 Once Daily | 0.2% CP-690,550 Once Daily | 0.02% CP-690,550 Once Daily | Placebo Once Daily | 2% CP-690,550 Twice Daily | 0.2% CP-690,550 Twice Daily | 0.02% CP-690,550 Twice Daily | Placebo Twice Daily
Number analyzed (Participants) | 4 | 3 | 4 | 1 | 9 | 6 | 11 | 2
ng/mg | 3.4145 (2.9877) | 2.2320 (2.7257) | 0.3242 (0.6343) | 0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable | 8.2810 (10.270) | 0.2957 (0.3675) | 0.0847 (0.1252) | 0 (NA) — Standard deviation was not estimable as only 2 participants were evaluable.

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | 2% CP-690,550 Once Daily | 0.2% CP-690,550 Once Daily | 0.02% CP-690,550 Once Daily | Placebo Once Daily | 2% CP-690,550 Twice Daily | 0.2% CP-690,550 Twice Daily | 0.02% CP-690,550 Twice Daily | Placebo Twice Daily
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/8 | 0/4 | 0/17 | 0/17 | 0/15 | 0/8
Other Adverse Events (participants affected / at risk) | 4/6 | 2/6 | 5/8 | 3/4 | 6/17 | 11/17 | 7/15 | 4/8
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2% CP-690,550 Once Daily (N=6) | 0.2% CP-690,550 Once Daily (N=6) | 0.02% CP-690,550 Once Daily (N=8) | Placebo Once Daily (N=4) | 2% CP-690,550 Twice Daily (N=17) | 0.2% CP-690,550 Twice Daily (N=17) | 0.02% CP-690,550 Twice Daily (N=15) | Placebo Twice Daily (N=8)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Application site irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Application site pruritus (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 2 | 0 | 0 | 1 | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.